CLINICAL TRIAL: NCT04946539
Title: Value of Ultrasonographic Enthesitis Assessment in Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Gunay ER, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 83045809-604.01.02
Record Dates: First submitted 2021-06-22; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Spondyloarthritis; Enthesitis
MeSH Terms: conditions — Spondylarthritis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spondyloarthritis
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Enthesitis assessment via ultrasonography

SUMMARY:
The aim of the study is to determine how valuable ultrasonographic enthesitis to asssess disease activity, functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Spondyloarthritis patients that fulfill 2009 ASAS criteria

Exclusion Criteria:

* history of elbow, ankle or knee surgery, local injection at the examination sites within the six weeks, peripheral neuropathy, infection and wound at examination site

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Spondyloarthritis
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Disease activity, | between November 2016 and January 2017
  BASDAI (Bath Ankylosing Spondylitis Disease Activity Index), minimum value 0, maximum value 10, higher scores mean a worse outcome
Disease activity, | between November 2016 and January 2017
  Ankylosing Spondylitis Disease Activity Score (ASDAS). It is calculated by adding CRP (ASDAS-CRP) or ESR (ASDAS-ESR). there is no spesific minimal and maximum value because it depends on CRP or ESR value. Higher scores mean a worse outcome
functionality | between November 2016 and January 2017
  Bath Ankylosing Spondylitis Functionality Index (BASFI). Minimal values 0, maximum value 100. Higher scores mean a worse outcome
to measure quality of life | between November 2016 and January 2017
  Short Form - 12 (SF-12). minimum value 0 maximum value 100. higher scores mean a worse outcome
to measure quality of life | between November 2016 and January 2017
  Ankylosing Spondylitis Quality of Life (ASQoL). minimum value 0 maximum value 18. Higher scores mean a worse outcome